CLINICAL TRIAL: NCT05572372
Title: Psychological Treatment of Hypersexuality: a Clinical Trial With Acceptance and Commitment Therapy
Brief Title: Effects of an ACT-based Psychological Treatment in Patients With Hypersexuality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Collaborators: apoyopositivo.org (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIPI/21/003
Record Dates: First submitted 2022-09-12; First posted 2022-10-07 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Compulsive Sexual Behavior; Hypersexuality
MeSH Terms: conditions — Compulsive Sexual Behavior Disorder | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ACT group (Experimental): Psychological intervention will consist in an 8-session individual on line-delivered ACT-based treatment.
  Interventions: Behavioral: Acceptance and Commitment Therapy

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — The aim of the intervention was to increase psychological flexibility. Therapeutic methods focused on values clarification, cognitive defusion, self-as-context, acceptance, commited action and flexible attention to present moment.

SUMMARY:
Investigation of the efficacy of Acceptance and Commitment Therapy (ACT) for the psychological treatment of hypersexuality.

DETAILED DESCRIPTION:
After being informed about the study, all patients giving written informed consent will be assessed to determine eligibility for study entry.

Patients who meet eligibility requirements will receive psychological intervention consisting in an 8-session individual on line-delivered ACT-based treatment.

The participants will be assessed through self-report instruments before and after treatment and at 3 months follow-up.

The clinical trial will not include a control group.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years-old
* Spanish speaking
* having had a sexual relationship in the last year
* significant score on the HBI Inventory (of 53 or more)
* at least 6 months of problematic pornography use or sexual practices
* clinically significant discomfort related to sexual practices
* degree of interference in his/her life of sexual practices greater than or equal to 5 out of 10
* at least one failure in his attempts to change his sexual life
* desire to improve/reduce excessive sexual behaviour

Exclusion Criteria:

* practicing meditation at least once a week in the last three months
* receiving psychological or psychopharmacological treatment
* intellectual disability
* substance dependence (use not associated with sex)
* personality disorder or other serious or chronic mental disorder diagnosed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-01-08 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Hypersexual Behavior Inventory (HBI) | Change from Baseline Hypersexuality at 5 months
  The Hypersexual Behavior Inventory is a 19-item, seven-point Likert-type scale. Scores range between 19 and 95. Higher scores indicate higher levels of Hypersexuality and worse outcome. García-Barba et al. (2020) consider the presence of a problem of hypersexuality when the score is equal or higher than 53.

SECONDARY OUTCOMES:
Change in Acceptance and Action Questionnaire (AAQ-II) | Change from Baseline psychological inflexibilty at 5 months
  Acceptance and Action Questionnaire assesses psychological inflexibility. It is a 7-item, seven-point Likert-type scale. Scores range between 7 and 49. Higher scores indicate higher levels of psychological inflexibility and worse outcome.
Change in Cognitive Fusion Questionnaire (CFQ) | Change from Baseline cognitive fusion at 5 months
  Cognitive Fusion Questionnaire assesses cognitive fusion. It is a 7-item, seven-point Likert-type scale. Scores range between 7 and 49. Higher the score in the questionnaire, the higher the tendency to believe the literal content of private events (higher levels of cognitive fusion and worse outcome).
Change in Scale of Body Connection (SBC) | Change from Baseline body awareness at 5 months
  Scale of Body Connection assesses Body Awareness (the capacity to be aware of body states, processes and actions, paying attention to the internal experience of the body) and Bodily Dissociation (avoidance of body experiences). It is a 20-item, 7-point Likert-type scale. Scores in Body Awareness scale range between 0 and 48. Higher scores indicate higher levels of body awareness and better outcome. Scores in Bodily Dissociation scale range between 0 and 32. Higher scores indicate higher levels of bodily dissociation and worse outcome.
Change in Mindful Attention Awareness Scale (MAAS) | Change from Baseline mindufullness skills at 5 months
  Mindful Attention Awareness Scale assesses mindfulness skills. It is a 15-item 6-point scale. Scores range between 1 and 6. Higher scores indicate a higher degree of attention to the present moment and a better outcome.
Change in The New Sexual Satisfaction Scale-short form (NSSS-S) | Change from Baseline sexual satisfaction at 5 months
  he New Sexual Satisfaction Scale assesses sexual satisfaction. It is a 12-item, 7-point Likert-type scale. Scores range between 12 and 60. Higher scores indicate a higher degree of sexual satisfaction and a better outcome.
Change in Intensity of cravings subjective scale | Through study completion, an average of 5 months
  Global self-assessment of intensity of cravings VAS-ratings. Scores range from 0 = very low intensity to 10 = very high intensity. Higher scores indicate higher levels of intensity of cravings and worse outcome.
Change in Interference of cravings subjective scale | Through study completion, an average of 5 months
  Global self-assessment of interference of cravings VAS-ratings. Scores range from 0 = very low interference to 10 = very high interference. Higher scores indicate higher levels of interference of cravings and worse outcome.
Change in Time spent planning or practicing sex per week | Through study completion, an average of 5 months
  Self-monitoring: Time spent (hours) planning or practicing sex during last week. Higher number of hours indicate worse outcome.
Change in number of sexual encounters per week | Through study completion, an average of 5 months
  Self-monitoring: Number of sexual encounters during last week. Higher number of sexual encounters indicate worse outcome.
Change in Frequency of chemsex encounters per week | Through study completion, an average of 5 months
  Self-monitoring: Frequency of practicing chemsex during last week. Higher number of chemsex encounters indicate worse outcome.
Change in number of different sexual partners per week | Through study completion, an average of 5 months
  Self-monitoring: Number of different sexual partners during last week. Higher number of different sexual partners indicate worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Montesinos, Ph.D., Principal Investigator — Universidad Europea de Madrid
Locations (1):
- Universidad Europea de Madrid, Villaviciosa de Odón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-08): https://cdn.clinicaltrials.gov/large-docs/72/NCT05572372/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-08): https://cdn.clinicaltrials.gov/large-docs/72/NCT05572372/ICF_001.pdf